CLINICAL TRIAL: NCT07308028
Title: Postural and Shoulder Function Norms Among Normal-Weight Children in Saudi Arabia: A Comparative Study With Obese School-Aged Peers
Brief Title: Postural and Shoulder Function Norms
Status: Completed | Type: Observational
Sponsor: Lincoln University College (Other)
Responsible Party: Principal Investigator, ALZAIDANI ABDULAZIZ ATIAH A, doctor, Lincoln University College
Other Study IDs: LUCMalaysia2
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Normal
Keywords: body mass index, isometric strength, range of motion, shoulder posture, school children.

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: forward head posture angle — angle between 2 lines; first line passing through tragus of the ear and seventh cervical vertebrae, the second line is horizontal line passing through seventh cervical vertebrae

SUMMARY:
Musculoskeletal development during childhood is influenced by several factors, including age, body composition, and physical activity. However, normative data regarding shoulder joint parameters and upper body posture among school-aged children in Saudi Arabia are lacking, particularly in relation to body mass index (BMI).

Objective: This study aims to establish normative reference values for shoulder joint mobility and upper body postural alignment in Saudi male school children, and to investigate the influence of BMI and age on these musculoskeletal parameters.

This study will provide foundational normative data for shoulder and upper body posture among school-aged children in Saudi Arabia and clarify the musculoskeletal impact of excess weight. The findings will support early screening and intervention strategies in pediatric populations.

DETAILED DESCRIPTION:
A cross-sectional analytical study will be conducted among 384 Saudi male students, aged 6 to 17 years, recruited from six randomly selected schools in the western region of Saudi Arabia. Participants will be stratified by BMI categories (normal, overweight, and obese) and age groups. Outcome measures will include forward head posture angle, shoulder slope angle, scapular downward rotation, and dorsal kyphosis. Other assessments will comprise shoulder pain intensity, functional disability, shoulder range of motion, and isometric strength. Descriptive statistics will be used to summarize demographic and clinical characteristics. A factorial multivariate analysis of variance (MANOVA) will be performed to assess the influence of BMI and age on the musculoskeletal parameters. Additionally, odds ratios (ORs) will be calculated to determine the association between obesity and postural abnormalities. Data will be analyzed using SPSS software version 26), with a significance level set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Saudi male students, aged 6 to 17 years

Exclusion Criteria:

* shoulder injuries previous shoulder surgery scoliosis

Ages: 6 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: 384 Saudi male students, aged 6 to 17 years, recruited from six randomly selected schools in the western region of Saudi Arabia. Participants will be stratified by BMI categories (normal, overweight, and obese) and age groups.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
shoulder pain intensity | one month
  measured on pain scale (visual analogue scale) from 0 (no pain ) to 10 (untolerable pain)

SECONDARY OUTCOMES:
functional disability | one month
  functional disability measured using shoulder disability index where higher scores indicates more disability

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Medical Complex, Ta'if, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided